CLINICAL TRIAL: NCT00829114
Title: Interactions Between Antiretrovirals and Combined Oral Contraceptive Pills
Brief Title: Interactions Between Antiretrovirals (ARVs) and Combined Oral Contraceptives (COCs)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Makerere University (Other); RHRU National Office, University of Witwatersand, Johannesburg (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10079
Record Dates: First submitted 2009-01-16; First posted 2009-01-26 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: HIV/AIDS; HIV Infections
Keywords: AE; AIDS; ALT; ART; AST; DCF; DMC; FDA; GCP; HB sAg; ICH; IND; IRB; IU; mg; mm3; PCR; SAE; ULN; WB; COC; Combined Oral Contraceptives
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): ART/COC group
  Interventions: Drug: ETHINYL ESTRADIOL AND LEVOGESTREL
- 2 (Active Comparator): COC group
  Interventions: Drug: ETHINYL ESTRADIOL AND LEVOGESTREL

INTERVENTIONS:
Drug: ETHINYL ESTRADIOL AND LEVOGESTREL — 30 MCG OF ETHINYL ESTRADIOL AND 150 MCG LEVOGESTREL
  Arms: 1
Drug: ETHINYL ESTRADIOL AND LEVOGESTREL — 30 MCG OF ETHINYL ESTRADIOL AND 150 MCG LEVOGESTREL
  Arms: 2

SUMMARY:
Non-randomized, comparative study (1:1 allocation) to study interactions between nevirapine-containing antiretroviral therapies and combined oral contraceptive pills.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent
* Willing to take COCs and follow all study requirements
* Has regular menstrual cycles every 21-35 days (when not taking hormonal contraception)
* Last menstrual period (LMP) <35 days before study entry
* Has body mass index of 18-30
* Negative urine pregnancy test as enrollment
* Documented HIV-1 infection
* On nevirapine-containing ART for at least three months (ART group only)
* CD4 cell count of greater than or equal to 350 (for non-ARV group only)
* Currently sexually active and plans to stay sexually active for the next 6 months

Exclusion Criteria:

* Medical contraindications to COC use
* Recent pregnancy (within 3 months)
* Has breastfed in last 3 months
* Last pregnancy was ectpoic
* Has been sterilized
* Has had any of the following conditions since last pregnancy, or since menarche if never pregnant:

Pelvic Inflammatory disease Diagnosis of infertility

* Has had DMPA within 6 months or NET injectable within 3 months of study entry (or has had no menses since last injection regardless of its timing)
* has taken other hormonal therapies besides COCs (e.g., combined injectables, progestin implants or intrauterine systems, progestin-only contraceptive pills, medroxyprogesterone acetate, hormone replacement therapy) within 30 days of study entry
* Has an acute infection or other opportunistic diseases requiring therapy within 14 days before enrollment
* Has active drug or alcohol use that, in the opinion of the investigator, would interfere with adherence to study requirements
* Has taken any prohibited medication within 30 days before study entry
* Has chronic diarrhea, malabsorption or inability to maintain an adequate oral intake
* Has any condition (social or medical) which in the opinion of the investigator would make study participation unsafe or complicate data interpretation

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 370 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Ovulation as determined by weekly blood progesterone (P) measurement | 2 months

SECONDARY OUTCOMES:
Pregnancy as detected by monthly urine pregnancy testing | 6 months
Adverse events (AE) recording | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Nanda, MD, Principal Investigator — FHI 360; Vera Halpern, MD, Principal Investigator — FHI 360
Locations (2):
- , RHRU National Office, University of Witwatersand, Esselent Saint Hillbrow, Johannesburg, South Africa
- Makerere University Medical School, Mulago Hospital, Department of Obstetrics and Gynecology, Kampala, Kampala, Uganda

REFERENCES:
- [Derived] Nanda K, Delany-Moretlwe S, Dube K, Lendvay A, Kwok C, Molife L, Nakubulwa S, Edward VA, Mpairwe B, Mirembe FM. Nevirapine-based antiretroviral therapy does not reduce oral contraceptive effectiveness. AIDS. 2013 Oct;27 Suppl 1:S17-25. doi: 10.1097/QAD.0000000000000050. PMID 24088680